CLINICAL TRIAL: NCT05915689
Title: Comparative Effects of Myofascial Arm Pull and Post Isometric Relaxation Techniques on Pain, Range of Motion and Functional Disability in Adhesive Capsulitis
Brief Title: Comparative Effects of Myofascial Arm Pull and Post Isometric Relaxation Techniques in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/23/0125
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis, Pain, Shoulder, Joint Range of Motion
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial arm pull technique (Experimental): subjects in this group will be treated with myofascial arm pull technique
  Interventions: Other: Myofascial arm pull technique
- Post Isomeric relaxation technique (Experimental): subjects in this group will be treated with post isometric relaxation technique
  Interventions: Other: post isometric relaxation technique

INTERVENTIONS:
Other: Myofascial arm pull technique — patient in supine position move the arm passively in abduction to the restricted barrier and pull the arm only enough traction was used to counterbalance the weight of the patient's arm. Stretch was hold until the fibers were released, and then, stretch was given again by increasing traction. This sequence was repeated until an end feel was reached. same procedure for flexion and scapular protraction and Horizontal-adduction. Repetition will be 4-5 reps. per set, 3 times per week for 18 sessions.
  Arms: Myofascial arm pull technique
Other: post isometric relaxation technique — The therapist stood in front of the patient, then placed one hand over the top of the subject's involved shoulder. The therapist cups the gleno humeral joint to palpate for motion and the subjects are directed to press the elbow towards therapist hand for shoulder abduction, internal rotation and external rotation. Muscle energy technique was applied for five repetitions per set, five sets per session, one session per day, three days a week for six weeks with each repetition maintained for the duration of 7-10 second
  Arms: Post Isomeric relaxation technique

SUMMARY:
Adhesive capsulitis is defined as a condition characterized by pain and stiffness in shoulder which results in both active and passive movement loss. The purpose of this study is to investigate the effects of shoulder directed treatment approach using Myofascial arm pull technique on the pain, range of motion and quality of life in patients with adhesive capsulitis and compare its effectiveness with Post Isometric Relaxation technique.

DETAILED DESCRIPTION:
Frozen shoulder is a common debilitating disorder characterized by shoulder pain and progressive loss of shoulder movement. Frozen shoulder is frequently associated with other systemic conditions or occurs following periods of immobilization, and has a protracted clinical course, which can be frustrating for patients as well as health-care professionals .Loyd define secondary frozen shoulder as a condition resulting from painful spasm on shoulder which causes activity limitation and dependency on opposite arm. In general population, the prevalence rate of frozen shoulder is around 2% to 5% and it ranges from 11% to 30% in diabetic population. Women are affected more than male and approx. 70% cases of frozen shoulder are on female. Among all frozen shoulder cases; around 20% to 30% patients develop frozen shoulder on opposite shoulder. Most of the frozen shoulder cases develop on non dominant shoulder. Adhesive Capsulitis of Shoulder is seen commonly at age of 40-65 years. Traditionally, FS has been regarded as a self-limiting and benign disease with complete recovery of pain and ROM. However, this condition can sometimes last for years. In one study, 50% of patients were still experiencing pain or stiffness of the shoulder at a mean of 7 years from the onset of the condition, although only 11% reported functional limitation. Different Physical therapy interventions used in patients with frozen shoulder frequently include modalities, manual techniques, and therapeutic exercise. Exercises given in the treatment of adhesive capsulitis consists of active ROM, Codman's exercise, wall walks, shoulder wheel, pulley, active and passive stretching, and rotator cuff and scapular strengthening exercises, METs, Gong mobilization, Mulligan mobilization. Many strategies have been employed in clinical practice to improve range and strength in prior research. There are limited studies regarding comparisons between the effects of myofascial arm pull and post isometric relaxation techniques that give the evidence of improving end painful ranges of adhesive capsulitis for long term effect. This study will be conducted to check the positive effect of myofascial arm pull technique and post isometric relaxation to increase end range in adhesive capsulitis. The literature review was conducted using different databases and the eleven selected articles fulfilled the criteria and included in research. Conclusion: Addition of Myofascial release technique and post isometric relaxation technique both as an adjunct to conventional treatment will have better benefits and faster recovery in patients with frozen shoulder but there are limited studies about the comparison of myofascial arm pull and post isometric relaxation techniques on pain, range of motion and quality of life in adhesive capsulitis. I will conduct this study to determine which technique is better to gain painful end ranges in adhesive capsulitis. So that this study will provide different treatment strategies for frozen shoulder to improve end painful ranges.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral frozen shoulder
* male and female
* Age between 40 and 60
* grade 2 frozen shoulder with pain lasting more than three month;
* capsular pattern of shoulder( External rotation, Abduction, Internal rotation)

Exclusion Criteria:

* Acute inflammation
* Subjects with systemic disease
* Dislocation and fracture in and around the shoulder,
* Rheumatoid arthritis
* History of Subjects with diabetes mellitus, osteoporosis or malignancies in shoulder region
* Past surgery around shoulder

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks
  An NPRS is described as an 11-point scale with scores from 0 to 10 and anchors of 0 = no pain and 10 = worst possible pain Numeric Rating Scale (NPRS) is most frequently used instruments to measure pain intensity in cervical spine. The 11-point numeric with 0 representing No pain, 1-3 representing Mild Pain (nagging, annoying, interfering little with ADLs), 4-6 representing Moderate Pains (interferes significantly with ADLs), 7-10 representing Sever Pain (disabling, unable to perform ADLs)
SPADI(shoulder pain and disability index) | 6 weeks
  The questionnaire consists of 13 items grouped into pain and disability subscales, the questions starting with "How severe is your pain." and "How much difficulty do you have.", respectively. Items mainly deal with various activities of daily living (ADL) that may or may not be problematic to the patient. Items are rated on visual analogue scales to produce a score for each subscale, and the means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst)

SECONDARY OUTCOMES:
Universal Goniometer | 6 weeks
  The universal mechanical goniometer (Plastic Goniometer-360 Degree Head - 12 inch arms) is a high-resolution plastic goniometer that permits observation of the axis of motion and ROM of the joint being measured The goniometer generally consists of a stationary arm, movable arm and a fulcrum. The circular or semi-circular portion is the centerpiece, which is the body of goniometer with a protractor printed on its face and the fulcrum of movable arm at its center. Generally, the fulcrum of the goniometer is placed over the center of a joint during measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Hafeez, PhD*, Principal Investigator — Riphah International University Lahore Campus
Locations (1):
- Hafeez clinic, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rangan A, Brealey SD, Keding A, Corbacho B, Northgraves M, Kottam L, Goodchild L, Srikesavan C, Rex S, Charalambous CP, Hanchard N, Armstrong A, Brooksbank A, Carr A, Cooper C, Dias JJ, Donnelly I, Hewitt C, Lamb SE, McDaid C, Richardson G, Rodgers S, Sharp E, Spencer S, Torgerson D, Toye F; UK FROST Study Group. Management of adults with primary frozen shoulder in secondary care (UK FROST): a multicentre, pragmatic, three-arm, superiority randomised clinical trial. Lancet. 2020 Oct 3;396(10256):977-989. doi: 10.1016/S0140-6736(20)31965-6. PMID 33010843
- [Background] Cho CH, Bae KC, Kim DH. Treatment Strategy for Frozen Shoulder. Clin Orthop Surg. 2019 Sep;11(3):249-257. doi: 10.4055/cios.2019.11.3.249. Epub 2019 Aug 12. PMID 31475043
- [Background] Tedla JS, Sangadala DR. Proprioceptive neuromuscular facilitation techniques in adhesive capsulitis: a systematic review and meta-analysis. J Musculoskelet Neuronal Interact. 2019 Dec 1;19(4):482-491. PMID 31789299
- [Background] Razzaq A, Nadeem RD, Akhtar M, Ghazanfar M, Aslam N, Nawaz S. Comparing the effects of muscle energy technique and mulligan mobilization with movements on pain, range of motion, and disability in adhesive capsulitis. J Pak Med Assoc. 2022 Jan;72(1):13-16. doi: 10.47391/JPMA.1360. PMID 35099430
- [Background] Duzgun I, Turgut E, Eraslan L, Elbasan B, Oskay D, Atay OA. Which method for frozen shoulder mobilization: manual posterior capsule stretching or scapular mobilization? J Musculoskelet Neuronal Interact. 2019 Sep 1;19(3):311-316. PMID 31475938
- [Background] Cohen C, Tortato S, Silva OBS, Leal MF, Ejnisman B, Faloppa F. Association between Frozen Shoulder and Thyroid Diseases: Strengthening the Evidences. Rev Bras Ortop (Sao Paulo). 2020 Aug;55(4):483-489. doi: 10.1055/s-0039-3402476. Epub 2020 Apr 6. PMID 32904783